CLINICAL TRIAL: NCT00931710
Title: A 12-week Multicenter, Randomized, Double-blind, Parallel-group, Active-control Study to Evaluate the Antihypertensive Efficacy and Safety of Valsartan/Amlodipine-based Regimen Versus a Losartan-based Regimen in Patients With Stage 2 Systolic Hypertension
Brief Title: Valsartan/Amlodipine As Compared to Losartan Treatment in Stage 2 Systolic Hypertension
Acronym: EXALT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVEA489AUS01
Record Dates: First submitted 2009-07-01; First posted 2009-07-02 (Estimated); Results first posted 2011-02-04 (Estimated); Last update posted 2011-03-07 (Estimated); Status verified 2011-03

CONDITIONS: Stage 2 Systolic Hypertension
Keywords: Hypertension; combination therapy; valsartan; cardiovascular diseases
MeSH Terms: conditions — Isolated Systolic Hypertension; Hypertension; Cardiovascular Diseases | interventions — Valsartan; Amlodipine; Hydrochlorothiazide; Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Valsartan/amlodipine/HCTZ (Experimental): Valsartan/amlodipine-based regimen: at randomization (Visit 3) patients were treated with valsartan/amlodipine 160/5 mg for 3 weeks, followed by a forced titration at Visit 4 (Week 3) to valsartan/amlodipine/HCTZ 160/5/25 mg for 3 weeks, and a second forced titration at Visit 5 (Week 6) to valsartan/amlodipine/HCTZ 320/10/25 mg for the remaining 6 weeks of the study.
  Interventions: Drug: valsartan, amlodipine, HCTZ
- Losartan/HCTZ (Active Comparator): Losartan-based regimen: at randomization (Visit 3) patients were treated with losartan 100 mg for 3 weeks, followed by a forced titration at Visit 4 (Week 3) to losartan/HCTZ 100/25 mg. At Visit 5 (Week 6) patients were switched to valsartan/amlodipine/HCTZ 160/5/25 mg for 3 weeks and, at Visit 6 (Week 9), patients were force titrated to valsartan/amlodipine/HCTZ 320/10/25 mg for the final 3 weeks of the study.
  Interventions: Drug: Losartan, HCTZ followed by valsartan, amlodipine, HCTZ

INTERVENTIONS:
Drug: valsartan, amlodipine, HCTZ — combination Valsartan/amlodipine160/5 mg tablet for 3 weeks; Valsartan/amlodipine 160/5mg tablet +HCTZ 25 mg capsule for 3 weeks; valsartan/amlodipine 320/10 mg tablet + HCTZ 25mg capsule for remainder (6 weeks) of the study
  Arms: Valsartan/amlodipine/HCTZ
Drug: Losartan, HCTZ followed by valsartan, amlodipine, HCTZ — losartan 100mg capsule for 3 weeks; losartan 100mg capsule +HCTZ 25 mg capsule for 3 weeks; Valsartan/amlodipine 160/5mg tablet +HCTZ 25 mg capsule for 3 weeks; valsartan/amlodipine 320/10 mg tablet + HCTZ 25mg capsule for remainder (3 weeks) of the study
  Arms: Losartan/HCTZ

SUMMARY:
This study will compare the antihypertensive efficacy and safety of a valsartan/amlodipine-based treatment with a losartan-based treatment in patients with Stage 2 systolic hypertension (high blood pressure, mean systolic blood pressure greater than 160 and less than 200 mmHg).

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatient of 18 years of age or greater
* Stage 2 systolic hypertension defined as office Mean Sitting Systolic blood pressure (MSSBP) greater than or equal to 160 and < 200 mmHg at randomization
* Patients who were able to participate in the study, and who gave written informed consent before any study assessment was performed.

Exclusion Criteria:

* Office systolic blood pressure >200 and/or mean sitting diastolic blood pressure (MSDBP) greater than or equal to 110 mmHg at Visit 1.
* Use of four (4) or more antihypertensive medications within 30 days of Visit 1.
* Refractory hypertension, defined as blood pressure >140/90 mmHg while taking three (3) drugs at the maximum dose of each drug, one of which must be a diuretic. (Therapy with a fixed-dose combination of two active medications represents two drugs).
* Inability to safely discontinue all antihypertensive medications for 1-2 weeks prior to randomization.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Actual)
Dates: Start 2009-07; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — 862-778-8300
Locations (1):
- sites in USA, East Hanover, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Losartan/HCTZ: Losartan-based regimen: at randomization (Visit 3) patients were treated with losartan 100 mg for 3 weeks, followed by a forced titration at Visit 4 (Week 3) to losartan/HCTZ 100/25 mg. At Visit 5 (Week 6) patients were switched to valsartan/amlodipine/HCTZ 160/5/25 mg for 3 weeks and, at Visit 6 (Week 9), patients were force-titrated to valsartan/amlodipine/HCTZ 320/10/25 mg for the final 3 weeks of the study.
Period: Overall Study
Arm/Group | Valsartan/Amlodipine/HCTZ | Losartan/HCTZ
Started | 241 | 247
Completed | 207 | 209
Not Completed | 34 | 38
Not completed — Adverse Event | 16 | 10
Not completed — Abnormal test procedure results | 2 | 0
Not completed — Unsatisfactory therapeutic effects | 5 | 12
Not completed — Patient withdrew consent | 4 | 9
Not completed — Lost to Follow-up | 6 | 5
Not completed — Protocol deviation | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Valsartan/Amlodipine/HCTZ | Losartan/HCTZ | Total
Number analyzed (Participants) | 241 | 247 | 488
Age Continuous [Mean (Standard Deviation); unit: years] | 55.0 (9.83) | 57.1 (9.69) | 56.1 (9.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 111 | 213
  Male | 139 | 136 | 275

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Sitting Systolic Blood Pressure After 6 Weeks
Description: To compare the change from baseline in mean sitting systolic blood pressure (MSSBP) after 6 weeks of valsartan/amlodipine-based regimen with a losartan-based regimen in patients with Stage 2 systolic hypertension.
Time Frame: Baseline to Week 6
Population: Full Analysis Set (FAS). Last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Valsartan/Amlodipine/HCTZ | Losartan/HCTZ
Number analyzed (Participants) | 241 | 247
mmHg
  Baseline | 166.8 (7.03) | 168.5 (9.03)
  Week 6 | 135.5 (16.26) | 142.5 (18.89)
  Change from Baseline to Week 6 | -31.3 (15.87) | -26.0 (16.62)

2. Secondary Outcome: Change in Mean Sitting Diastolic Blood Pressure After 6 Weeks
Description: To compare the change from baseline in mean sitting diastolic blood pressure (MSDBP) after 6 weeks of valsartan/amlodipine-based regimen with losartan-based regimen in patients with Stage 2 systolic hypertension.
Time Frame: Baseline to Week 6
Population: Full Analysis Set (FAS). Last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Valsartan/Amlodipine/HCTZ | Losartan/HCTZ
Number analyzed (Participants) | 241 | 247
mmHg
  Baseline | 98.6 (7.71) | 97.6 (7.88)
  Week 6 | 85.1 (10.05) | 88.5 (11.36)
  Change from Baseline to Week 6 | -13.6 (9.48) | -9.1 (10.03)

3. Secondary Outcome: Cumulative Percentage of Patients Achieving Blood Pressure Control
Description: To compare the percentage of patients achieving blood pressure control (defined as patients achieving MSSBP < 140 mmHg and MSDBP < 90 mmHg) after 3 and 6 weeks of valsartan/amlodipine-based regimen with losartan-based regimen in patients with Stage 2 systolic hypertension.
Time Frame: 3 and 6 weeks
Population: Full Analysis Set (FAS).
Measure: Number; unit: cumulative percentage of patients
Arm/Group | Valsartan/Amlodipine/HCTZ | Losartan/HCTZ
Number analyzed (Participants) | 241 | 247
cumulative percentage of patients
  Week 3 | 30.5 | 15.3
  Week 6 | 61.5 | 47.1

4. Secondary Outcome: Cumulative Percentage of Treatment Responders
Description: To compare the percentage of treatment responders (defined as patients with MSSBP < 140 mmHg or demonstrating a decrease from baseline of ≥ 20 mmHg) after 3 and 6 weeks of valsartan/amlodipine-based regimen with losartan-based regimen in patients with Stage 2 systolic hypertension.
Time Frame: 3 and 6 weeks
Population: Full Analysis Set (FAS).
Measure: Number; unit: Cumulative percentage of responders
Arm/Group | Valsartan/Amlodipine/HCTZ | Losartan/HCTZ
Number analyzed (Participants) | 241 | 247
Cumulative percentage of responders
  Week 3 | 65.3 | 34.3
  Week 6 | 87.0 | 71.5

5. Secondary Outcome: Change in Mean Sitting Systolic and Diastolic Blood Pressure After 12 Weeks
Description: To compare the change from baseline in MSSBP and MSDBP after 12 weeks of valsartan/amlodipine-based regimen with losartan-based regimen in patients with Stage 2 systolic hypertension.
Time Frame: Baseline to week 12
Population: Full Analysis Set (FAS). Last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Valsartan/Amlodipine/HCTZ | Losartan/HCTZ
Number analyzed (Participants) | 241 | 247
mmHg
  Baseline MSSBP | 166.8 (7.03) | 168.5 (9.03)
  Week 12 MSSBP | 130.8 (16.22) | 134.3 (19.41)
  Change in MSSBP from baseline to Week 12 | -36.0 (16.08) | -34.2 (17.69)
  Baseline MSDBP | 98.6 (7.71) | 97.6 (7.88)
  Week 12 MSDBP | 82.5 (10.18) | 82.5 (11.43)
  Change in MSDBP from baseline to Week 12 | -16.1 (9.91) | -15.1 (10.57)

6. Secondary Outcome: Cumulative Percentage of Patients With Incidence of Peripheral Edema Before or at the Corresponding Visit
Description: To assess the incidence of peripheral edema occurring with valsartan/amlodipine-based regimen versus losartan-based regimen in patients with Stage 2 systolic hypertension.
Time Frame: 3, 6, 9 and 12 weeks
Population: Full Analysis Set (FAS).
Measure: Number; unit: cumulative percentage of patients
Arm/Group | Valsartan/Amlodipine/HCTZ | Losartan/HCTZ
Number analyzed (Participants) | 241 | 247
cumulative percentage of patients
  Week 3 | 0.8 | 0.8
  Week 6 | 0.8 | 0.8
  Week 9 | 1.3 | 0.8
  Week 12 | 2.9 | 4.5

ADVERSE EVENTS:
Groups:
- Valsartan / Amlodipine / HCTZ: Valsartan / amlodipine / HCTZ
- Losartan / HCTZ: Losartan / HCTZ
Arm/Group | Valsartan / Amlodipine / HCTZ | Losartan / HCTZ
Serious Adverse Events (participants affected / at risk) | 1/241 | 2/247
Other Adverse Events (participants affected / at risk) | 13/241 | 8/247
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Valsartan / Amlodipine / HCTZ (N=241) | Losartan / HCTZ (N=247)
Non-cardiac chest pain (General disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Valsartan / Amlodipine / HCTZ (N=241) | Losartan / HCTZ (N=247)
Dizziness (Nervous system disorders) | 13 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.